CLINICAL TRIAL: NCT05182879
Title: Evaluation of Frail Elderly in Ambulatory Primary Care
Acronym: EPAFRA
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2016_23; 2016-A01750-51 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2021-12-22; First posted 2022-01-10 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Frailty
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Assessement with GERONTOPOLE scale — The practitionner assesses the frailty of the elderly outpatient with the GERONTOPOLE scale and compares it with the "évaluation gériatrique standardisée" (GDS)

SUMMARY:
Evaluate the sensitivity of the GERONTOPOLE scale, used by general practitioners in primary care outpatients for the diagnosis of frailty in non-dependent people more than 65 years old, using as reference the "évaluation gériatrique standardisée clinique" (EGS)

ELIGIBILITY:
Inclusion Criteria:

* Independent patients

Exclusion Criteria:

* Dependent outpatient, assessed with a "activity of daily living" (ADL) score < 6/6
* outpatient with occuring severe health episode less than a month before inclusion

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly independent population
Sampling Method: Probability Sample
Enrollment: 740 (Estimated)
Dates: Start 2019-02-12 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
assess the sensitivity of the GERONTOPOLE scale | 2 years
  by practitionner

CONTACTS AND LOCATIONS:
Overall Officials: Nassir MESSAADI, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- CHU Lille, Lille, Nord, France

IPD SHARING:
Plan to Share IPD: No